CLINICAL TRIAL: NCT03486509
Title: Phase II Study of Afatinib Plus Chemotherapy in Patients With Esophageal and Lung Squamous Cell Carcinoma
Brief Title: Afatinib Plus Chemotherapy Against Esophageal or Lung Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSWOG201702
Record Dates: First submitted 2017-12-18; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2017-12

CONDITIONS: Squamous Cell Carcinoma
Keywords: afatinib
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Afatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- afatinib 40mg bid plus chemotherapy (Experimental): afatinib 40mg bid po plus chemotherapy
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — afatinb 40mg po bid

SUMMARY:
As a 2nd generation EGFR-TKI that irreversibly binds to EGFR receptors, afatinib is currently recommended as the standard first-line treatment for EGFR mutation-positive lung cancer, and clinical studies are also being actively conducted in other types of carcinomas characterized by EGFR gene mutation and overexpression.

The overall results from previous studies of gefitinib and erlotinib as EGFR TKIs , as well as from preceding studies of afatinib - a 2nd generation EGFR TKI - suggest the possibility of an effective therapy in esophageal cancer or squmaous lung cancer. In this phase II trial, afatinib shall be administered to patients with squamous cell carcinoma of esophagus or lung squamous cell carcinoma to evaluate its effects and toxicity. Also, biomarkers to predict responses to afatinib shall be explored through further studies.

DETAILED DESCRIPTION:
As a 2nd generation EGFR-TKI that irreversibly binds to EGFR receptors, In a phase III study LUX-lung 8 in patients with squamous lung cancer, afatinib monotherapy showed longer progression-free disease survival than erlotinib therapy. afatinib is currently recommended as the standard first-line treatment for EGFR mutation-positive lung cancer, and clinical studies are also being actively conducted in other types of carcinomas characterized by EGFR gene mutation and overexpression. Thirty (30) solid cancer patients were included in a phase I trial of afatinib, and of them, a patient with esophageal cancer had partial response. Taken together, based upon the results from clinical trials of afatinib conducted so far, 7 out of 15 esophageal cancer patients achieved clinical responses of 3 months or longer.

Hence, the overall results from previous studies of gefitinib and erlotinib as EGFR TKIs and our study of dacomitinib, as well as from preceding studies of afatinib - a 2nd generation EGFR TKI - suggest the possibility of an effective therapy in esophageal cancer or squmaous lung cancer. In this phase II trial, afatinib shall be administered to patients with squamous cell carcinoma of esophagus or lung squamous cell carcinoma to evaluate its effects and toxicity. Also, biomarkers to predict responses to afatinib shall be explored through further studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must understand the rigors of the study and provide written informed consent and HIPAA authorization prior to initiation of any study procedures
* Life expectancy > 10 months
* Karnofsky Performance Status ≥ 70
* Diagnosis of histological or cytologically confirmed squamous lung cancer or esophageal squamous cancer,
* Age ≥ 18 years
* Adequate organ and bone marrow function, defined as: Bone marrow: absolute neutrophil count (ANC) ≥ 1.5 x 109/L; hemoglobin > 9 g/dL; platelets > 100 x 109/L Renal: creatinine clearance ≥ 50 mL/min (calculated according to Cockroft and Gault) or creatinine ≤ 1.5 mg/dL Hepatic: bilirubin ≤ 1.5 x the upper limit of normal (ULN); aspartate transaminases (AST/SGOT) and alanine transaminases (ALT/SGPT) ≤ 2.5 x ULN (or ≤ 5 x ULN if due to underlying liver metastases); internation normalized value for prothrombin time (INR) ≤ 1.5 x ULN (except in the case of anticoagulation therapy), albumin ≥ 2.0
* Good medical candidate for and willing to undergo a biopsy or surgical procedure to obtain tissue, which may or may not be part of the patient's routine care for their malignancy.

Exclusion Criteria:

* Poor compliance, reluctant to undergo research medication, or follow-up.
* Tumor inaccessible for biopsy
* It is currently included in clinical trials of other drugs, or at the same time, into other medical studies that are considered incompatible with the study.
* It has a history of other cancers, unless the cancer is completely relieved and has not been treated for more than 3 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
PFS | through study completion, an average of 2 year
  Progression-Free-Survival

SECONDARY OUTCOMES:
ORR | through study completion, an average of 2 year
  objective response rate

OTHER OUTCOMES:
adverse events | through study completion, an average of 2 year
  the Common Terminology Criteria for Adverse Events ver. 4.0

IPD SHARING:
Plan to Share IPD: Undecided